CLINICAL TRIAL: NCT05510414
Title: Evaluation of a Psychological Capital Intervention to Alleviate Burnout and Regulate Immunity Among Oncology Nurses: a Randomized Controlled Trial
Brief Title: Evaluation of a Psychological Capital Intervention to Alleviate Burnout and Regulate Immunity Among Oncology Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, professor, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PCI burnout
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Burnout; Psychological
Keywords: Burnout; oncology nurses; positive psychology capital intervention; immune variables
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: The intervention program was taught by experts with at least the title of deputy chief nurse who had been engaged in clinical psychological nursing for a long time. These teachers helped nurses with burnout to develop their own positive psychology, learn optimism, embrace hope, find available support systems and resources, plan their careers. Training took the form mainly of Balint groups, lectures, group discussions, video watching and outdoor development. Personalized counseling was provided to address specific psychological problems in individuals, in a way that ensured personal privacy. The intervention occurred as 12 sessions of 60 min each, twice a month, lasting altogether six months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI group (Experimental): intervention based on psychological capital model
  Interventions: Behavioral: psychological intervention based on psychological capital
- Control group (No Intervention): routine psychological counseling

INTERVENTIONS:
Behavioral: psychological intervention based on psychological capital — Psychological capital would be modified via various training programs in order to manage burnout among nurses. When the four core psychological resources are combined, they may form a higher-order construct that predicts attitudes and performance more strongly than any of the four components by themselves .
  Arms: PCI group

SUMMARY:
Burnout appears to be highly prevalent among oncology nurses, which was a problem not only for the nurses themselves but for the patients for whom they provide care. How to mitigate and prevent burnout and improve nursing performance outcomes is an urgent problem for nursing manager.

In a sample of 99 oncology nurses, immunological characteristics were compared to burnout scores. In a randomized trial, 90 oncology nurses suffering burnout were randomized to receive psychological capital intervention or routine psychological care. Participants were assessed before and after treatment using measures of burnout, psychological capital and immunological characteristics.

DETAILED DESCRIPTION:
Burnout appears to be highly prevalent among oncology nurses, which was a problem not only for the nurses themselves but for the patients for whom they provide care. And burnout-associated biomarkers remain controversial, and their potential roles in burnout are still unclear.

This study was a randomized controlled trial in which the independent variable was group psychological intervention, while the dependent variables were pre- and post-intervention scores on the Maslach burnout inventory and on the psychological capital scale, as well as values for various immunological indicators. In Stage 1 of the study, recruited subjects completed the psychological capital questionnaire and blood was sampled. In Stage 2, the research team administered a custom-designed psychological capital intervention (PCI) to part of the sample, while the other part received routine care . The PCI group received 1 h of counseling twice weekly for a total of 24 weeks in total. In Stage 3, the PCI and control groups completed the questionnaires again and provided blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were officially employed and licensed nurses who had been working in the cancer hospital for at least 2 years.

Exclusion Criteria:

* Subjects had recently suffered personal health problems or significant negative life events, such as the death or serious illness of a family member, or if they were on maternity leave or other types of leave from their nursing job.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
scores on Maslach Burnout Inventory-General Survey (MBI-GS) | baseline and 6 months
  change of the MBI scores, which ranges from 0 to 6, with higher scores indicating more severe burnout.

SECONDARY OUTCOMES:
scores on Positive psychological capital Questionnaire (PPQ), | baseline and 6 months
  change of the PPQ scores, , which ranges from 1 to 6, with higher scores indicating higher level of psychological capital.

CONTACTS AND LOCATIONS:
Overall Officials: Xue-Mei You, MD, Principal Investigator — Guangxi Medical University Cancer Hospital
Locations (1):
- Affiliated Tumor of Guangxi University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] An M, Shin ES, Choi MY, Lee Y, Hwang YY, Kim M. Positive Psychological Capital Mediates the Association between Burnout and Nursing Performance Outcomes among Hospital Nurses. Int J Environ Res Public Health. 2020 Aug 18;17(16):5988. doi: 10.3390/ijerph17165988. PMID 32824724
- [Background] Ciobanu AM, Damian AC, Neagu C. Association between burnout and immunological and endocrine alterations. Rom J Morphol Embryol. 2021 Jan-Mar;62(1):13-18. doi: 10.47162/RJME.62.1.02. PMID 34609405
- [Background] Luo YH, Li H, Plummer V, Cross WM, Lam L, Guo YF, Yin YZ, Zhang JP. An evaluation of a positive psychological intervention to reduce burnout among nurses. Arch Psychiatr Nurs. 2019 Dec;33(6):186-191. doi: 10.1016/j.apnu.2019.08.004. Epub 2019 Aug 19. PMID 31753226